CLINICAL TRIAL: NCT07324681
Title: Evaluation of Irisin Levels in Adult Patients With Forearm Fractures Undergoing Surgery With Infraclavicular Block and General Anesthesia
Brief Title: Evaluation of Irisin Levels in Adult Forearm Fracture Surgery Under Infraclavicular Block and General Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TABED 1-25-1099
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Inflamation; Healing; Angiogenesis
Keywords: irisin; infraclavicular block; forearm fracture
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (GA) Group (Active Comparator): Adult patients undergoing elective forearm fracture surgery under general anesthesia. Standard noninvasive monitoring will be used and perioperative hemodynamic variables and analgesic use will be recorded. Blood samples for serum irisin will be collected preoperatively, at 30 minutes postoperatively, and at 24 hours postoperatively.
  Interventions: Procedure: General Anesthesia (GA)
- Infraclavicular Block (ICB) Group (Experimental): Adult patients undergoing elective forearm fracture surgery with an ultrasound-guided infraclavicular brachial plexus block performed approximately 1 hour before surgery under monitored conditions. Standard noninvasive monitoring will be used; perioperative hemodynamic variables and analgesic use will be recorded. Blood samples for serum irisin will be collected preoperatively, at 30 minutes postoperatively, and at 24 hours postoperatively.
  Interventions: Procedure: Infraclavicular Brachial Plexus Blocks

INTERVENTIONS:
Procedure: General Anesthesia (GA) — General anesthesia administered according to institutional routine; anesthetic drugs and doses will be recorded.
  Arms: General Anesthesia (GA) Group
Procedure: Infraclavicular Brachial Plexus Blocks — Ultrasound-guided infraclavicular block performed preoperatively; details of technique, local anesthetic drugs and doses will be recorded.
  Arms: Infraclavicular Block (ICB) Group

SUMMARY:
This randomized prospective study evaluates the effect of general anesthesia versus infraclavicular nerve block on perioperative serum irisin levels in adults undergoing forearm fracture surgery. Irisin levels will be measured preoperatively, at 30 minutes postoperatively, and at 24 hours postoperatively. The association between irisin changes and fracture healing will be explored as a secondary outcome.

DETAILED DESCRIPTION:
Forearm fractures are common injuries in adults and frequently require surgical intervention due to instability and displacement. Postoperative recovery quality and fracture healing are influenced by multiple factors, including the type of anesthesia administered during surgery. However, the biochemical and metabolic effects of different anesthesia techniques on bone healing remain insufficiently explored.

Irisin is a myokine derived from the cleavage of fibronectin type III domain-containing protein 5 (FNDC5) and plays a significant role in muscle-bone crosstalk. Experimental and clinical studies have demonstrated that irisin promotes osteoblast differentiation, inhibits osteocyte apoptosis, and contributes to bone homeostasis and fracture healing. Despite its potential importance, the relationship between anesthesia techniques and perioperative irisin levels has not been previously investigated.

This single-center, randomized, prospective clinical trial aims to compare the effects of general anesthesia and infraclavicular brachial plexus block on perioperative serum irisin levels in adult patients undergoing elective forearm fracture surgery. Patients aged 18-65 years with American Society of Anesthesiologists (ASA) physical status I-III will be randomly assigned to one of two groups: general anesthesia (Group G) or infraclavicular block (Group B).

Serum irisin levels will be measured at three time points: preoperatively, 30 minutes postoperatively, and 24 hours postoperatively. In addition to biochemical outcomes, intraoperative hemodynamic parameters (heart rate, blood pressure, oxygen saturation), analgesic consumption, and demographic data will be recorded. Postoperative radiographs will be evaluated to monitor fracture healing and callus formation, which will be analyzed as a secondary outcome in relation to changes in irisin levels.

The primary outcome of the study is the comparison of perioperative changes in serum irisin levels between the two anesthesia techniques. Secondary outcomes include the relationship between irisin level changes and radiological fracture healing, as well as differences in perioperative physiological stress responses.

This study aims to improve understanding of the metabolic and biochemical effects of anesthesia techniques on bone healing. The findings may contribute to the selection of anesthesia methods that minimize physiological stress and potentially enhance postoperative recovery and fracture healing in patients undergoing forearm fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years

Scheduled for elective forearm fracture surgery

Planned to receive either general anesthesia or infraclavicular brachial plexus block

American Society of Anesthesiologists (ASA) physical status I-III

Able to provide written and verbal informed consent

Exclusion Criteria:

* Age <18 years or >65 years

Emergency surgery

Refusal or inability to provide informed consent

ASA physical status IV or V

Known bone diseases or metabolic bone disorders

Multiple trauma or associated organ injury

Inability to mobilize

Morbid obesity (BMI >40 kg/m²)

Renal failure

Hepatic failure

Neurological deficits or sequelae

Contraindication or allergy to any anesthetic agents used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Irisin Levels | Preoperative (baseline), 30 minutes postoperatively, and 24 hours postoperatively
  Serum irisin levels (ng/dL) will be measured to evaluate the effect of anesthesia type on perioperative irisin response. Blood samples will be collected at three time points: preoperatively (baseline), 30 minutes postoperatively, and 24 hours postoperatively. Changes in irisin levels will be compared between the general anesthesia group and the infraclavicular block group.

SECONDARY OUTCOMES:
Radiological Fracture Healing and Callus Formation | Postoperative follow-up period (up to 6 months)
  Postoperative radiographs will be evaluated to assess fracture healing and callus formation. Radiological findings will be analyzed in relation to perioperative changes in serum irisin levels to explore a potential association between irisin response and fracture healing.

CONTACTS AND LOCATIONS:
Overall Officials: sumru sekerci, professor, Study Director — Ankara Bilkent City Hospital Department of Anesthesiology and Reanimation, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient privacy concerns and institutional data protection policies. De-identified aggregate data will be reported in publications.

REFERENCES:
- [Result] Bostrom P, Wu J, Jedrychowski MP, Korde A, Ye L, Lo JC, Rasbach KA, Bostrom EA, Choi JH, Long JZ, Kajimura S, Zingaretti MC, Vind BF, Tu H, Cinti S, Hojlund K, Gygi SP, Spiegelman BM. A PGC1-alpha-dependent myokine that drives brown-fat-like development of white fat and thermogenesis. Nature. 2012 Jan 11;481(7382):463-8. doi: 10.1038/nature10777. PMID 22237023